CLINICAL TRIAL: NCT03707262
Title: Donor Chimerism and Graft Survival Following Combined HLA-Identical Sibling Living Donor Kidney and Hematopoietic Stem Cell Transplantation Utilizing a Conditioning Regimen of Total Lymphoid Irradiation and Rabbit Anti-Thymocyte Globulin
Brief Title: Study of Combined Kidney and Blood Stem Cell Transplant From a Brother or Sister Donor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeffrey Veale, MD (Other)
Collaborators: OneLegacy Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Jeffrey Veale, MD, Professor, David Geffen School of Medicine, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLA-Match Tolerance
Record Dates: First submitted 2018-08-01; First posted 2018-10-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Renal Transplant Rejection; Tolerance; Kidney Transplant
Keywords: Tolerance; Kidney Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Donor CD34+ and CD3+ cell infusion (Experimental): The investigational products are (1) an intravenous infusion of granulocyte colony-stimulating factor (GCSF)-mobilized, Miltenyi-enriched CD34+ cells (≥ 5 million cells per kilogram) followed by (2) an infusion of CD3+ cells (5 million cells per kilogram) from an HLA-identical sibling living donor.
  The cells are infused around Day 11 post-transplant after the following pre-conditioning regimen:
  1. 5 doses of rATG (1.5 mg/kg IV per day for 5 days, starting on the day of transplant)
  2. 10 doses of TLI (120 centigray [cGY] x 10 fractions, starting the day after transplant)
  Interventions: Biological: Donor CD34+ and CD3+ cells

INTERVENTIONS:
Biological: Donor CD34+ and CD3+ cells — Infusion of GCSF-mobilized, Miltenyi-enriched CD34+ hematopoietic stem/progenitor cells (HSPCs) (≥ 5 million cells/kg) and CD3+ cells (5 million cells/kg) from an HLA-identical sibling living donor, following pre-conditioning regimen of rATG and TLI.

SUMMARY:
The purpose of this study is to find out if an investigational treatment will allow kidney transplant recipients to better accept their new kidney and stop immunosuppressive medicines. This study is for kidney transplant recipients who receive a kidney from a sibling donor.

The investigational treatment is started after kidney transplant. It begins with a regimen of a drug called rabbit anti-thymocyte globulin (rATG) combined with radiation therapy (known as total lymphoid irradiation, or TLI) to the lymph nodes and spleen. This is followed by an infusion of blood stem cells, which will be donated by the same sibling who donated their kidney. Researchers think that this treatment allows immune cells from the donor and recipient to live side by side, a condition referred to as "mixed chimerism." Mixed chimerism may help create a state of "tolerance" in kidney transplant recipients in which all immunosuppressive medications can be stopped without rejection of the transplanted kidney.

This study will test whether (1) the investigational treatment will allow patients to stop immunosuppressive medications after their kidney transplant and (2) if the treatment impacts the rate of kidney rejection and the side effects of immunosuppressive medications.

DETAILED DESCRIPTION:
In spite of the pronounced benefit of kidney transplantation in prolonging survival and improving the quality of life of patients with end stage renal disease, it is still hampered by the risk of graft rejection and the need for lifelong immunosuppression. Researchers have sought to circumvent these challenges through the use of combined kidney and hematopoietic stem cell transplantation to induce immune tolerance. This study will build upon published reports showing favorable results for the TLI/rATG regimen in HLA-matched living donor transplant recipients. The investigators seek to confirm that patients treated with total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG) followed by human leukocyte antigen (HLA)-identical donor hematopoietic progenitor cell transplant can be withdrawn from immunosuppressive drugs while maintaining normal renal function after renal transplantation. At serial time points, (1) graft function will be monitored, (2) chimerism will be measured in recipient white blood cell subsets, and (3) protocol biopsies of the graft will be obtained. An attempt will be made to discontinue tacrolimus at 12 months if the following conditions are met: (1) chimerism (defined as ≥5% donor type cells among the T cells, B cells, Natural Killer [NK] cells, and granulocytes) is detectable for at least 180 days after CD34+ and CD3+ cell infusion, (2) stable graft function without clinical rejection episodes is maintained, (3) there is lack of histologic rejection on protocol biopsies, and (4) there is no evidence of graft vs. host disease (GVHD). Recipients in the proposed study will be given a target dose of ≥ 5 x106 CD34+ cells/kg and 5x106 CD3+ cells/kg with the goal of achieving durable mixed chimerism.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Males and females ages 18 years and older receiving living donor kidney transplant from an HLA-identical sibling at UCLA Medical Center.
2. Agrees to participate in the study and is able to give informed consent.
3. Resides or is willing to stay within 3 hours distance from UCLA Medical Center by ground transportation for the first three to six months of the trial at the physician's discretion.
4. Meets institutional criteria for kidney and HSPC transplant.
5. No known contraindication to administration of rATG or radiation.
6. If patient is a female of reproductive potential (i.e., no documented absence of ovaries or uterus, history of tubal ligation, or post-menopausal status) patient must be confirmed not pregnant by a serum or urine pregnancy test) and must agree to practice a reliable form of contraception including hormonal treatments, barrier methods or intrauterine device for at least 12 months post-transplant. Karnofsky Performance Score ≥ 70.
7. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 40% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
8. Adequate pulmonary function defined as FVC and DLCO of greater than or equal to 50% of predicted.
9. Adequate liver function defined as total bilirubin ≤ 1.5 times the upper limit of normal and AST/ALT ≤ 2.0 times the upper limit of normal.
10. Adequate social support based on evaluation by the UCLA renal transplant team licensed clinical social worker.

Recipient Exclusion Criteria:

1. Donor is identical twin.
2. ABO incompatibility with donor.
3. Previous solid organ transplant
4. Multi-organ transplantation
5. Previous treatment with rATG or a known allergy to rabbit proteins
6. History of active malignancy within the past 5 years with the exception of non-melanomatous skin cancer.

   a. History of another primary malignancy except for: i. Malignancy treated with curative intent and with no known active disease >2 years before the first dose of study treatment and of low potential risk for recurrence ii. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease iii. Very low risk and low risk cancer adequately treated or on active surveillance b. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, and DCIS)
7. Pregnant (confirmed by urine or serum pregnancy test) or lactating.
8. Leukopenia (with a white blood cell count < 3,000/ µL) or thrombocytopenia (with a platelet count < 100,000/ µL).
9. Active bacterial, fungal, mycobacterial or viral infection (including active hepatitis B and/or C).
10. Positive HLA DSA
11. Seropositivity for HIV 1, HIV 2, HTLVI, HTLV II
12. Active West Nile Virus infection
13. Renal disease with high risk of recurrence (i.e., focal segmental glomerulosclerosis).
14. Advanced hepatic fibrosis or cirrhosis secondary to hepatitis B and/or C diagnosis.
15. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia; active extra-renal autoimmune disease requiring immunosuppression.
16. Active extra-renal autoimmune disease requiring immunosuppression.
17. Neuropsychiatric illness that precludes the ability to give informed consent and/or places the patient as high risk for non-compliance with the safety monitoring requirements of the study.
18. May not have received other immunosuppressive medications, including but not limited to alemtuzumab, belatacept, sirlolimus, everolimus, azathioprine, basiliximab, and eculizumab within six months of the study treatment. Use of corticosteroids prescribed for a time-limited indication (</= 4 weeks) and stopped at least 4 weeks before the kidney transplant is acceptable.
19. May not have received immunotherapy drugs such as immune checkpoint inhibitors (e.g. pembrolizumab, nivolumab, and ipilimumab), tumor necrosis factor inhibitors, rituximab, and interleukin-2 within six months of the study treatment.
20. Current or active abuse of alcohol and/or drugs within last 6 months.
21. BMI 40 or greater.

Donor Inclusion Criteria:

1. HLA-identical sibling on high-resolution HLA typing who is ≥18 years of age.
2. Meets institutional criteria for living kidney and allogeneic HSPC transplant donation.
3. Medically fit to tolerate peripheral blood apheresis, including weighing ≥110 pounds, hemoglobin ≥ 11 g/dL, white blood cell count ≥ 3,000/µL, and platelets ≥120,000/µL.
4. Normal serum chemistry and coagulation studies; or, if abnormal, the differences are not considered clinically significant.

Donor Exclusion Criteria:

1. Recipient is identical twin.
2. ABO incompatibility with recipient.
3. Medically unfit to tolerate peripheral blood apheresis (small body size, poor vascular access, not a suitable candidate for placement of a central catheter, etc.).
4. Pregnant (confirmed by urine or serum pregnancy test) or lactating.
5. Seropositivity for HIV 1, HIV 2, HTLV I, HTLV II
6. Active West Nile Virus infection
7. Active bacterial, fungal, mycobacterial or viral infection (including active hepatitis B and/or C)
8. Psychiatric, addictive, neurological, or other disorder that compromises ability to give true informed consent for participation in this study

   1. History of active malignancy within the past 5 years with the exception:Adequately managed malignancy within the past two years with low risk of recurrence may be acceptable as per clinician discretion
   2. Adequately managed non-melanoma skin cancer
   3. Adequately managed carcinoma in situ e.g., cervical cancer in situ, and DCIS
9. No current or recent use of oral anti-coagulants. (For the purpose of this study, recent is defined as less than 60 days prior to apheresis.). Note: Use of aspirin and non-steroidal anti-inflammatory drugs, for pain and inflammation management purposes, are permitted to enroll in the study, but these drugs must be stopped 14 days prior to apheresis, however subjects who are taking aspirin for its anti-platelet/anti-thrombotic effect, are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Withdrawal from immunosuppressive drugs | 12 months post-kidney transplant
  Percentage of subjects free from all immunosuppressive drugs at 12 months after kidney transplantation.

SECONDARY OUTCOMES:
Graft rejection | 48 months post-kidney transplant
  Percentage of patients with graft rejection within 48 months post-transplant defined as (1) meets Banff criteria for rejection either on protocol biopsy or biopsy performed to confirm clinical suspicion of rejection or (2) clinical suspicion of rejection demonstrating response to corticosteroids in absence of biopsy when confirmatory biopsy contraindicated or declined.
Time to graft rejection | 48 months post-kidney transplant
  Time to graft rejection
Graft failure | 48 months post-kidney transplant
  Percentage of patients with graft failure as determined by return to dialysis and/or re-transplantation.
Time to graft failure | 48 months post-kidney transplant
  Time to graft failure
Survival | 12, 24, 36, and 48 months post-kidney transplant
  Percentage of subjects alive at 12, 24, 36, and 48 months post-kidney transplant
Time to death | 48 months post-kidney transplant
  Time to death (months post-transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Veale, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
N/A, undecided